CLINICAL TRIAL: NCT05466344
Title: Assessment of the Condylar Response of Mini-plate Anchored Rigid Fixed Functional Appliance Versus Dentally Anchored Semi-rigid One; A Randomized Clinical Trial
Brief Title: the Condylar Response of Mini-plate Anchored Rigid Fixed Functional Appliance Versus Dentally Anchored Semi-rigid One
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mahmoud M. Fathy Aboelmahasen, Clinical professor of orthodontics - Faculty of dental medicine, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 603/307
Record Dates: First submitted 2022-07-16; First posted 2022-07-20 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Class II Malocclusion
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Intervention Model Description: Participants will be selected based on the following inclusion criteria:
  1. Skeletal class 2 malocclusion due to mandibular retrusion with increased overjet (SNA= 82±4, ANB=≥4°). With agefrom 18 to 25 years.
  2. Mandibular arch with minimum (up to 4mm) or no crowding.
  3. All permanent teeth are erupted (3rd molar not included).
  4. Good oral and general health.
  5. No systemic disease or regular medication that could interfere and/or affect orthodontic teeth movement.
  6. No previous orthodontic treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herbst Group (Active Comparator): Include ten young adult orthodontic patients who are treated by using fixed orthodontic appliances followed by the type IV Herbst appliance (mini plate anchored appliance). The age of patients will be (18-20y).
  Interventions: Device: Herbst Group
- TFBC Group (Active Comparator): Include ten young adult orthodontic patients who are treated by using fixed orthodontic appliances followed by the Twin Force Bite Corrector appliance (dentally anchored appliance). The age of patients will be (18-20y).
  Interventions: Device: TFBC Group

INTERVENTIONS:
Device: Herbst Group — 1. Two mini plates are chosen, the last hole in every plate is used to solder the ball housing of type IV Herbst appliance.
  2. The two mini plates are placed bilateral at the mandibular symphysis and fixed by at least 3 screws, the surgical wound is sutured leaving an extended part of the plate in the oral cavity which contain the soldered ball housing.
  3. The surgical wound is left for 2 weeks for proper soft tissue healing, in the meantime separation in the arch, band placement on the first premolar and molar bilateral followed by impression for construction of the upper Herbst splint.
  4. Cementation of upper Herbst splint with connecting the telescopic piston through fitting of the plunger into the tube bilaterally.
  5. When reactivation of the telescopic piston is needed, extension rings are used.
  Other Names: Group I
  Arms: Herbst Group
Device: TFBC Group — 1. The patients will be treated by fixed orthodontic appliance with using series of orthodontic NiTi arch wires for levelling and alignment.
  2. Installation of series of orthodontic stainless steel arch wires until 0.0019 x 0.0025 inch for both arches.
  3. Installation of the Twin Force Bite Corrector appliance for 4 to 6 months.
  4. Using of class ΙΙ intra-oral elastics for both sides for 2 to 3 months.
  5. Finally follow finishing steps for each patient.
  Other Names: Group II
  Arms: TFBC Group

SUMMARY:
This study will be directed to evaluate The effect of two different types of fixed functional appliances on the temporomandibular joint.

Study design:

Prospective randomized clinical study.

Study setting and population:

This study will be conducted on twenty orthodontic patients. The number of patients was dependent on a power study.

Sample size calculation was based on the observed average effect size derived from previous article addressing "the effect of skeletally anchored Forsus FRD using miniplates for the treatment of Class II malocclusion

DETAILED DESCRIPTION:
Participants will be selected based on the following inclusion criteria:

1. Skeletal class 2 malocclusion due to mandibular retrusion with increased overjet (SNA= 82±4, ANB=≥4°).
2. Mandibular arch with minimum (up to 4mm) or no crowding.
3. All permanent teeth are erupted (3rd molar not included).
4. Good oral and general health.
5. No systemic disease or regular medication that could interfere and/or affect orthodontic teeth movement.
6. No previous orthodontic treatment.

outcomes measures:

1. primary outcome: comparison of condylar volume of Herbst group versus TFBC group.
2. secondary outcome: Measurement of of condylar volume within each group (Herbst group and TFBC group)

Treatment steps:

As for Group Ι:

1. Two mini plates are chosen, the last hole in every plate is used to solder the ball housing of type IV Herbst appliance.
2. The two mini plates are placed bilateral at the mandibular symphysis and fixed by at least 3 screws, the surgical wound is sutured leaving an extended part of the plate in the oral cavity which contain the soldered ball housing.
3. The surgical wound is left for 2 weeks for proper soft tissue healing, in the meantime separation in the arch, band placement on the first premolar and molar bilateral followed by impression for construction of the upper Herbst splint.
4. Cementation of upper Herbst splint with connecting the telescopic piston through fitting of the plunger into the tube bilaterally.
5. When reactivation of the telescopic piston is needed, extension rings are used.

As for Group ΙΙ:

1. The patients will be treated by fixed orthodontic appliance with using series of orthodontic NiTi arch wires for levelling and alignment.
2. Installation of series of orthodontic stainless steel arch wires until 0.0019 x 0.0025 inch for both arches.
3. Installation of the Twin Force Bite Corrector appliance for 4 to 6 months.
4. Using of class ΙΙ intra-oral elastics for both sides for 2 to 3 months.
5. Finally follow finishing steps for each patient.

Observations:

Changes in the condylar volume and changes in position of the condyle in relation to glenoid fossa as a result of remodeling process before and after the fixed functional orthopedic treatment at each group.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be selected based on the following inclusion criteria:

  1. Skeletal class 2 malocclusion due to mandibular retrusion with increased overjet (SNA= 82±4, ANB=≥4°). With agefrom 18 to 25 years.
  2. Mandibular arch with minimum (up to 4mm) or no crowding.
  3. All permanent teeth are erupted (3rd molar not included).
  4. Good oral and general health.
  5. No systemic disease or regular medication that could interfere and/or affect orthodontic teeth movement.
  6. No previous orthodontic treatment.

Exclusion Criteria:

- 1. Patients with a blocked-out tooth that will not allow for placement of the bracket at the initial bonding appointment.

2. Patients with untreated decay or any endodontic lesions.

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
comparison of condylar volume of Herbst group versus TFBC group | nine months
  three dimensional automatic measurement of condylar volume as one unit by Romexis software

SECONDARY OUTCOMES:
Measurement of of condylar volume within each group (Herbst group and TFBC group) | nine months
  three dimensional automatic measurement of condylar volume as one unit by Romexis software

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Fathy, PHD, Principal Investigator — Clinical professor of orthodontics - Faculty of dental medicine - Al-Azhar university
Locations (1):
- Mahmoud Mohammad Fathy Abo - Elmahasen, Maadi, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No